CLINICAL TRIAL: NCT03003533
Title: Gene-transfer, Open-label, Dose-escalation Study of SPK-8011 [Adeno-associated Viral Vector With B-domain Deleted Human Factor VIII Gene] in Individuals With Hemophilia A
Brief Title: A Gene Transfer Study for Hemophilia A
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPK-8011-101
Record Dates: First submitted 2016-12-16; First posted 2016-12-28 (Estimated); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Hemophilia A
Keywords: Adeno-Associated Virus (AAV); Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Factor VIII (FVIII); Factor VIII (FVIII) Deficiency; Factor VIII (FVIII) Gene; Factor VIII (FVIII) Protein; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Gene Therapy; Gene Transfer; Hematologic Diseases; Hemorrhagic Disorders; Recombinant; Vector
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Hematologic Diseases; Hemorrhagic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SPK-8011 5x10^11 vg/kg (Experimental): Participants received a single intravenous (IV) infusion of SPK-8011 5x10^11 vector genomes per kilogram (vg/kg) body weight.
  Interventions: Genetic: SPK-8011
- SPK-8011 1x10^12 vg/kg (Experimental): Participants received a single IV infusion of SPK-8011 1x10^12 vg/kg.
  Interventions: Genetic: SPK-8011
- SPK-8011 2x10^12 vg/kg (Experimental): Participants received a single IV infusion of SPK-8011 2x10^12 vg/kg.
  Interventions: Genetic: SPK-8011
- SPK-8011 1.5x10^12 vg/kg (Experimental): Participants received a single IV infusion of SPK-8011 1.5x10^12 vg/kg.
  Interventions: Genetic: SPK-8011

INTERVENTIONS:
Genetic: SPK-8011 — A novel, bio-engineered, recombinant adeno-associated viral vector carrying human factor VIII gene

SUMMARY:
This clinical research study is being conducted by Spark Therapeutics, Inc. to determine the safety and efficacy of the factor VIII gene transfer treatment with SPK-8011 in individuals with hemophilia A.

DETAILED DESCRIPTION:
Hemophilia A is a condition in which blood is unable to clot effectively. It is caused by a mutation or deletion in the gene that is responsible for producing blood-clotting factor VIII protein. Individuals with hemophilia A suffer from repeated bleeding episodes, often into the joints, which can cause chronic joint disease and sometime results in death due to the inability of the blood to clot efficiently. This chronic joint disease can have significant physical, psychosocial, and quality-of-life effects, including financial burden. The current standard of care includes the use of factor-based therapies which are given either as prophylaxis or to treat bleeding, as well as new non-factor prophylaxis therapies.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18 years or older
* Confirmed diagnosis of hemophilia A as evidenced by their medical history with baseline FVIII activity levels <=2%
* Have received >150 exposure days (EDs) to FVIII concentrates or cryoprecipitate
* Have no prior history of allergic reaction to any FVIII product
* Have no measurable inhibitor against FVIII as assessed by the central laboratory and have no prior history of inhibitors to FVIII protein and no clinical signs or symptoms of decreased response to FVIII administration
* Agree to use reliable barrier contraception

Exclusion Criteria:

* Evidence of active hepatitis B or C
* Currently on antiviral therapy for hepatitis B or C
* Have significant underlying liver disease
* Have serological evidence* of HIV-1 or HIV-2 with CD4 counts ≤200/mm3 and who are on an antiretroviral drug regimen (* participants who are HIV+ and stable with CD4 count >200/mm3 and undetectable viral load are eligible to enroll)
* Have detectable antibodies reactive with AAV-Spark200 capsid
* Participated in a gene transfer trial within the last 52 weeks or in a clinical trial with an investigational product within the last 12 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Director, Study Director — Spark Therapeutics, Inc.
Locations (16):
- United States (11):
  - University of California Davis - Hemostasis and Thrombosis Center, Sacramento, California
  - University of Florida Health, Gainesville, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Weill Cornell Medicine-Comprehensive Center for Hemophilia and Coagulation Disorders, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Pennsylvania State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
- Australia (2):
  - Royal Prince Alfred Hosptial, Camperdown, New South Wales
  - The Alfred Hospital, Melbourne
- McMaster University Medical Centre and Juravinski Hospital, Hamilton, Ontario, Canada
- Chaim Sheba Center, Ramat Gan, Tel Hashomer, Israel
- Mahidol University - Ramathibody Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] George LA, Monahan PE, Eyster ME, Sullivan SK, Ragni MV, Croteau SE, Rasko JEJ, Recht M, Samelson-Jones BJ, MacDougall A, Jaworski K, Noble R, Curran M, Kuranda K, Mingozzi F, Chang T, Reape KZ, Anguela XM, High KA. Multiyear Factor VIII Expression after AAV Gene Transfer for Hemophilia A. N Engl J Med. 2021 Nov 18;385(21):1961-1973. doi: 10.1056/NEJMoa2104205. PMID 34788507
- [Derived] Ran G, Chen X, Xie Y, Zheng Q, Xie J, Yu C, Pittman N, Qi S, Yu FX, Agbandje-McKenna M, Srivastava A, Ling C. Site-Directed Mutagenesis Improves the Transduction Efficiency of Capsid Library-Derived Recombinant AAV Vectors. Mol Ther Methods Clin Dev. 2020 Mar 13;17:545-555. doi: 10.1016/j.omtm.2020.03.007. eCollection 2020 Jun 12. PMID 32258217

RESULTS

PARTICIPANT FLOW:
Groups:
- SPK-8011 5x10^11 vg/kg: Participants received a single intravenous infusion of SPK-8011 5x10^11 vector genomes per kilogram body weight (vg/kg).
- SPK-8011 1x10^12 vg/kg: Participants received a single intravenous infusion of SPK-8011 1x10^12 vg/kg.
- SPK-8011 2x10^12 vg/kg: Participants received a single intravenous infusion of SPK-8011 2x10^12 vg/kg.
- SPK-8011 1.5x10^12 vg/kg: Participants received a single intravenous infusion of SPK-8011 1.5x10^12 vg/kg.
Period: Overall Study
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Started | 2 | 3 | 9 | 11
Received at Least 1 Dose of Study Drug | 2 | 3 | 9 | 11
Completed | 2 | 3 | 9 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Groups:
- SPK-8011 5x10^11 vg/kg: Participants received a single intravenous infusion of SPK-8011 5x10^11 vg/kg.
- Total: Total of all reporting groups
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg | Total
Number analyzed (Participants) | 2 | 3 | 9 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 9 | 11 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 2 | 3 | 9 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 9 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 2 | 2 | 9 | 10 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as adverse events that result in death, are life-threatening, require inpatient hospitalization or prolongation of existing hospitalization, result in persistent or significant disability or incapacity, are a congenital anomaly or birth defect, or are an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE is defined as an AE with an onset date on or following SPK-8011 administration. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From date of first dose to Week 52/End of Study (EOS) Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
Participants | 2 | 3 | 9 | 11

2. Primary Outcome: Number of Participants Who Received Corticosteroids for Presumed Immune Response
Time Frame: Up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
Participants | 0 | 2 | 7 | 10

3. Primary Outcome: Peak Factor VIII (FVIII) Activity Levels Assessed by One-Stage Coagulation Assay (OSA)
Description: Median peak FVIII activity up to Week 52
Time Frame: Up to Week 52/EOS visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Median (Full Range); unit: percentage of normal activity
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
percentage of normal activity | 11.5 [11 to 12] | 20.0 [6 to 24] | 38.7 [7 to 209] | 55.1 [31 to 112]

4. Primary Outcome: Nominal FVIII Level by OSA at Week 52/EOS
Description: Steady-state FVIII activity measured by median FVIII levels at week 52 by OSA.
Time Frame: Up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of normal activity
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 6 | 11
percentage of normal activity | 5.4 [4.7 to 6.1] | 7.8 [3.0 to 13.9] | 8.4 [3.0 to 19.7] | 4.1 [3.0 to 11.9]

5. Primary Outcome: Spontaneous Bleeds Annualized Bleeding Rate
Time Frame: Week 5 up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Median (Inter-Quartile Range); unit: annualized number of bleeding events
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
annualized number of bleeding events | NA [NA to NA] — Median and IQR not calculable due to insufficient number of participants in the arm | 0.3 [0.2 to 0.6] | 0.0 [0.0 to 1.4] | 0.0 [0.0 to 0.7]

6. Primary Outcome: Total Annualized FVIII Infusion Rate
Time Frame: Week 5 up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Mean (Standard Deviation); unit: total annualized FVIII infusions
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
total annualized FVIII infusions | 0.3 (0.40) | 3.6 (3.18) | 7.4 (7.93) | 1.6 (1.81)

7. Secondary Outcome: Time to Achieve Peak FVIII Activity Level
Time Frame: Up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
days | 279.5 (58.69) | 141.0 (151.79) | 56.4 (19.84) | 54.6 (33.74)

8. Secondary Outcome: Number of Participants With Vector-shedding Confirmed Below Quantifiable Limits (BQL) of SPK-8011-101 in Bodily Fluids
Time Frame: Up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
Participants
  Peripheral blood mononuclear cells (PBMCs) | 2 | 3 | 9 | 11
  Saliva | 2 | 3 | 9 | 10
  Semen | 2 | 2 | 8 | 11
  Serum | 2 | 3 | 8 | 10
  Urine | 2 | 3 | 9 | 10

9. Secondary Outcome: Incidence of Immune Response to the BDD-hFVIII Transgene
Time Frame: Up to Week 52/EOS Visit
Population: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Measure: Count of Participants; unit: Participants
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
Number analyzed (Participants) | 2 | 3 | 9 | 11
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to Week 52
Description: The Full Analysis Set included all participants who received the infusion of SPK-8011.
Arm/Group | SPK-8011 5x10^11 vg/kg | SPK-8011 1x10^12 vg/kg | SPK-8011 2x10^12 vg/kg | SPK-8011 1.5x10^12 vg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 1/9 | 3/11
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 9/9 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPK-8011 5x10^11 vg/kg (N=2) | SPK-8011 1x10^12 vg/kg (N=3) | SPK-8011 2x10^12 vg/kg (N=9) | SPK-8011 1.5x10^12 vg/kg (N=11)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPK-8011 5x10^11 vg/kg (N=2) | SPK-8011 1x10^12 vg/kg (N=3) | SPK-8011 2x10^12 vg/kg (N=9) | SPK-8011 1.5x10^12 vg/kg (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Normocytic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1
Scleral Hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Gingival Discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Intestinal Mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Salivary Gland Mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Face Oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 3
Feeling Hot (General disorders) | 0 | 0 | 0 | 1
Feeling Jittery (General disorders) | 0 | 0 | 0 | 1
Generalised Oedema (General disorders) | 0 | 0 | 0 | 1
Hunger (General disorders) | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hyperplastic Cholecystopathy (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Allergy To Arthropod Sting (Immune system disorders) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 2 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 1
Dermatitis Infected (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Herpes Dermatitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 1 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Nail Infection (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2
Otitis Media Acute (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pulpitis Dental (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 4
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 1
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Animal Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chemical Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 5
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 1
Glycosylated Haemoglobin Increased (Investigations) | 0 | 1 | 0 | 0
Sars-Cov-2 Test Positive (Investigations) | 0 | 0 | 1 | 1
Transaminases Increased (Investigations) | 0 | 0 | 2 | 5
Weight Increased (Investigations) | 0 | 0 | 1 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Seronegative Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 4
Morton's Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 1
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 4
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
Testicular Disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1
Pharyngeal Swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT03003533/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03003533/SAP_001.pdf